CLINICAL TRIAL: NCT03809754
Title: Optical Coherence Tomography Guided Percutaneous Coronary Intervention for Drug-eluting In-stent Restenosis: A Prospective Registry Trial
Brief Title: Optical Coherence Tomography Guided Percutaneous Coronary Intervention for Drug-eluting In-stent Restenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yun Dai Chen, Professor, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Z171100001017158
Record Dates: First submitted 2019-01-15; First posted 2019-01-18 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: CHD - Coronary Heart Disease; Percutaneous Coronary Intervention; In-stent Restenosis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OCT-guided PCI (Experimental)
  Interventions: Procedure: Percutaneous Coronary Intervention under OCT
- Angiography-guided PCI (Sham Comparator)
  Interventions: Procedure: Percutaneous Coronary Intervention under Angiography

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention under OCT — After randomization, subjects receive primary PCI under the guiding of OCT
  Arms: OCT-guided PCI
Procedure: Percutaneous Coronary Intervention under Angiography — After randomization, subjects receive primary PCI under the guiding of angiography
  Arms: Angiography-guided PCI

SUMMARY:
This study is a prospective, registry trial aimed to compare the clinical and angiographic outcomes of OCT-guided and angiography-guided PCI in patients with coronary DES-ISR.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patients with angina or evidence of myocardial ischaemia
* Patients with restenotic lesions in a previously DES area of a coronary artery
* Patients suitable to receive any types of percutaneous coronary intervention (including balloon angioplasty and stent implantation)
* The stent diameter of DES-ISR is 2.5mm to 4.0mm
* Target lesion length < 30mm
* Target lesion stenosis ≥ 70% diameter stenosis on visual assessment, or ≥ 50% diameter stenosis and with evidence of myocardial ischaemia ischemic

Exclusion Criteria:

* Patients with acute myocardial infarction with 1 week
* Patients with evidence of extensive thrombosis in the target vessel
* Patients with left main coronary artery disease
* Patients with cardiogenic shock, left ventricular ejection fraction < 40%,significant renal dysfunction and severe heart valve disease
* Patients who had cerebral stroke within 6 months before PCI
* Patients with a life expectancy < 1 year
* Patients not able to adhere to follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
In-segment late loss at 9 months follow-up | 9 months

SECONDARY OUTCOMES:
Rates of acute success | 1 month
Rate of 9-month binary restenosis | 9 months
Number of Participants with target lesion failure (TLF) | 12 months
Rate of major adverse cardiovascular events | 12 months
Number of participants with all-cause death | 12 months
Rate of myocardial infarction | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yundai Chen, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Yundai Chen, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Han Y, Yuan X, Wang W, Wang N, Zhang Y, Jing J, Chen Y, Gao L. Clinical Significance of Optical Coherence Tomography-Guided Percutaneous Coronary Intervention for In-Stent Restenosis Within Drug-Eluting Stents: Impact on Patient Outcomes. J Am Heart Assoc. 2024 Nov 5;13(21):e033954. doi: 10.1161/JAHA.123.033954. Epub 2024 Nov 4. PMID 39494577